CLINICAL TRIAL: NCT05389852
Title: Analgesic Efficacy of Intravenous Dexmedetomidine for Supraclavicular Plexus Block: a Randomized Double-blinded Placebo Controlled Clinical Trial
Brief Title: Analgesic Efficacy of Intravenous Dexmedetomidine for Supraclavicular Plexus Block
Acronym: TwoDex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hôpital du Valais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hopitalduvalais
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-03

CONDITIONS: Surgery
Keywords: locoregional anesthesia; postoperative analgesia; hand surgery; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients undergoing forearm or hand surgery under supraclavicular brachial plexus block, receiving either additional intravenous dexmedetomidine or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: dexmedetomidine or placebo prepared by Lausanne University Hospital Pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous dexmedetomidine (Active Comparator): Patients will receive intravenous dexmedetomidine 1 mcg/kg just after the supraclavicular brachial plexus block is completed
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Patients will receive intravenous placebo (normal saline) just after the supraclavicular brachial plexus is completed
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — After completion of supraclavicular brachial plexus block patients will receive intravenous dexmedetomidine 1 mcg/kg
  Other Names: Dexdor

SUMMARY:
The goal of the study is to compare the duration of analgesia in patients undergoing forearm or hand surgery with a supraclavicular brachial plexus block, who receive either iv dexmedetomidine or placebo.

DETAILED DESCRIPTION:
Most surgical interventions on the forearm and the hand in Valais Hospital are performed under regional anesthesia. This ensures intraoperative patient comfort and reduces pain during the first 6 to 12 postoperative hours. A very common strategy to provide anesthesia of the arm is to inject local anesthetics in the region over the clavicle around the brachial plexus. This "supraclavicular brachial plexus block" is routinely performed in Valais Hospital and is always done under ultrasound guidance.

A drawback of locoregional anesthesia is the recurrence of pain once the effect of the block wears off after approximately 6 to 8 hours. This phenomenon is called rebound pain. It and can be very severe and debilitating, can significantly impact postoperative recovery and may also preclude ambulatory surgery as well as early mobilization and physiotherapy. Therefore, strategies that prolong the analgesic effect of locoregional anesthesia are warranted.

Dexmedetomidine is a selective α2-adrenoceptor agonists with sedative and analgesic properties. It has been shown to prolong the analgesic duration of local anesthetics when administered intravenously. However, the association of dexmedetomidine with long-acting local anesthetics for supraclavicular brachial plexus block has not been systematically investigated.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elbow, forearm or hand surgery under supraclavicular brachial plexus block Patients who are ASA physical status I-III

Exclusion criteria

* Patient refusal
* ASA physical status IV
* History of hypersensitivity or intolerance to dexmedetomidine
* History of hypersensitivity or intolerance to dexamethasone
* History of hypersensitivity or intolerance to local anesthetics
* History of recent (< 1 year) cerebrovascular insult
* Second or third degree heart block
* Uncontrolled hypotension
* Conditions contraindicating supraclavicular brachial plexus block: neurological deficit or neuropathy of the arm, severe hepatic dysfunction (Child B and C), coagulopathy, malignancy or infection in the area above the clavicle
* Chronic opioid use
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
duration of analgesia | 24 hours on day of surgery
  time in minutes from end of injection of local anesthetic till first analgesic request

SECONDARY OUTCOMES:
Duration of motor block | 24 hours on day of surgery
  time in minutes from completion of locoregional anesthesia and the moment the patient can again mobilize the arm
Duration of sensory block | 24 hours on day of surgery
  time in minutes from completion of locoregional anesthesia and the moment the patient regains sensation of the arm
Pain scores at rest | 4, 24, 48 hours postoperatively
  Pain scores at rest on numeric scale, 0=no pain at all to 10=worst pain imaginable
Pain scores on movement | 4, 24, 48 hours postoperatively
  Pain scores on movement, on numeric scale, 0=no pain at all to 10=worst pain imaginable
Cumulative amount of opiate analgesic medication consumed | 24, 48 hours postoperatively
  in intravenous morphine equivalents (mg)
Patient satisfaction | 7 days postoperatively
  on 4 point Likert scale: dissatisfied / neutral / satisfied / extremely satisfied
Total number of dexmedetomidine-related side effects | 24 hours postoperatively
  Total number of dexmedetomidine-related side effects, in particular bradycardia and hypotension
Dexmedetomidine-related side effects | 24 hours postoperatively
  Number and % of patients who experience at least one dexmedetomidine-related side effect
Opioid-related side effect | 24 hours postoperatively
  Number and % of patients who experience at least one opioid-related side effect

CONTACTS AND LOCATIONS:
Overall Officials: Sina Grape, MD, MBA, Principal Investigator — Valais Hospital
Locations (1):
- Hopital du Valais, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grape S, Andany A, Cibotto C, Berri L, Rossel JB, Albrecht E. Duration of analgesia after supraclavicular brachial plexus block with intravenous dexamethasone with or without dexmedetomidine: a randomised, placebo-controlled, triple-blind trial. Br J Anaesth. 2025 Dec 1:S0007-0912(25)00792-5. doi: 10.1016/j.bja.2025.10.049. Online ahead of print. PMID 41330797